CLINICAL TRIAL: NCT07393529
Title: A Pilot Randomized Controlled Trial of a Social Network Intervention for Older Patients With Cancer
Brief Title: A Pilot Randomized Controlled Trial of a Social Network Intervention
Acronym: SONATA 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UOCPC26005
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cancer; Older Adults (65 Years and Older); Social Networks
Keywords: geriatric oncology; social networks
MeSH Terms: interventions — zaleplon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SONATA Intervention (Experimental): Following randomization, patients assigned to SONATA will participate in up to six coaching sessions, delivered either in person or via Zoom over approximately six weeks.
  Interventions: Behavioral: SONATA
- Enhanced Usual Care (No Intervention): Patients randomized to enhanced usual care will receive standard educational materials within 4 weeks of randomization.

INTERVENTIONS:
Behavioral: SONATA — SONATA includes six evidence-based components to help patients: 1) identify and set personal goals to achieve well-being (goal-setting); 2) identify their social network (SN) members and map their SNs (network diagnostics); 3) engage key SN members to address their goals and needs (network engagement); 4) build channels for communication and collaboration with key SN members via in-person and virtual activities (opportunity creation); 5) communicate effectively with their key SN members, develop action plans, and provide support (skill building); and 6) engage in cycles of feedback to effectively respond to the patient's evolving needs.
  Arms: SONATA Intervention

SUMMARY:
This is a pilot randomized controlled trial to assess the feasibility, acceptability, appropriateness, and structure of the SONATA intervention. In addition, it will assess the preliminary efficacy of SONATA compared to enhanced usual care among 70 older adults with advanced cancer.

DETAILED DESCRIPTION:
Older adults (aged ≥65) with advanced cancer are living longer due to more effective treatments, but their median survival remains around one year. We have shown that this population experiences a high prevalence of aging-related conditions, including functional and cognitive impairments, as well as depressive and anxiety symptoms. These conditions heighten their vulnerability to treatment toxicities and increase their need for assistance with daily activities. Together, these challenges impair older adults' ability to manage their care (patient activation) and reduce their overall quality of life (QoL). Therefore, interventions are needed to increase patient activation and improve QoL in this vulnerable population.

Fostering supportive social networks (SNs) can help older adults navigate the burden of cancer and its treatments. SNs comprise individuals (e.g., family members and friends) connected by interpersonal relationships. SN members offer a range of support, including instrumental, emotional, and informational support. They play pivotal roles in clinical settings, particularly for older individuals with functional impairments. SN members attend clinic visits and advocate for patients, ensuring accurate exchange and filtering of information to align with patients' preferences. SN members also shape patients' identities, coping strategies, and disease understanding. The role of SNs becomes more prominent as older adults become more ill.

The SOcial Networks to Activate Teamwork & Alliance (SONATA) intervention was designed to harness the SNs to provide support to older adults with advanced cancer and increase patient activation and improve QoL. The objective of this study is to conduct a pilot randomized controlled trial assessing SONATA compared to enhanced usual care among 70 older adults with advanced cancer.

ELIGIBILITY:
Patients

Inclusion criteria:

* Age ≥65 years
* A diagnosis of advanced or likely incurable cancer, as determined by the primary oncologist
* Able to speak English
* Able to provide informed consent

Exclusion criteria:

* Any psychiatric or cognitive impairments interfering with participation as determined by the oncology team
* Unwilling to complete study procedures

Social Network Members (if available, for intervention arm only)

Inclusion criteria:

* Age ≥18 years
* Identified as an SN member by the patient in the intervention arm
* Able to speak English
* Able to provide informed consent

Exclusion criteria:

• Unwilling to complete study procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Study feasibility | From baseline to week 16
  Retention rate. Percentage of patients who complete at least three SONATA sessions and week 16 post-intervention assessments

SECONDARY OUTCOMES:
Emotional, social, and existential quality of life | From baseline to week 16
  14-item McGill QoL Questionnaire-Revised. A 14-item survey assessing quality of life. It has four subscales: Physical, Psychological, Existential, and Social. We will focus on Psychological, Existential, and Social subscales. Mean scores range from 0 to 10, higher scores are better
Patient Activation | From baseline to week 16.
  Patient Activation Measure. A 13-item survey to assess patient knowledge, skill, and confidence for self-management. Total scores range from 0 to 100, higher scores are better.
Autonomy, Competence, and Relatedness | From baseline to week 16
  Basic Psychological Need Satisfaction Scale. A 21-item survey to assess the degree to which people feel satisfaction of these three needs - autonomy, competence, and connectedness. Total scores range fom 21 to 147, higher scores are better.
Social Support | From baseline to week 16
  Medical Outcomes Study-Social Support Survey. A 19-item survey to assess four domains of emotional/informational support, instrumental support, positive social interaction, and affection. Total scores range from 0-100, higher scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Permission will also be asked on the consent form for the use of patient and social network (SN) data for future research not described in this consent. In addition, permission will be asked from patients and SN members to share de-identified transcripts from recordings for future research not described in the consent.
Supporting Information: Study Protocol
Time Frame: All study data will be kept for a period of 7 years after the date of study closure.

REFERENCES:
- [Background] Kehoe L, Sanapala C, DiGiovanni G, Yousefi-Nooraie R, Yilmaz S, Bauer J, Loh KP, Norton S, Duberstein P, Kamen C, Gilmore N, Gudina A, Kleckner A, Mohile S, Epstein RM. Older adults with advanced cancer are selective in sharing and seeking information with social networks. Patient Educ Couns. 2022 Oct;105(10):3116-3122. doi: 10.1016/j.pec.2022.06.005. Epub 2022 Jun 9. PMID 35717349
- [Background] Yu V, Yilmaz S, Freitag J, Loh KP, Kehoe L, Digiovanni G, Bauer J, Sanapala C, Epstein RM, Yousefi-Nooraie R, Mohile S. The role of social networks in prognostic understanding of older adults with advanced cancer. Patient Educ Couns. 2023 Jan;106:135-141. doi: 10.1016/j.pec.2022.10.009. Epub 2022 Oct 15. PMID 36270857